CLINICAL TRIAL: NCT03851679
Title: Pulmonary Echography and BNP Value Pre- and Post- Elective Cesarean Section in Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: University of Udine (Other)
Responsible Party: Principal Investigator, Bove, Professor, University of Udine
Other Study IDs: BNP and pulmonary echography
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Pregnancy Related
Keywords: pulmonary echography; B-Type natriuretic peptide; Spinal anesthesia
MeSH Terms: interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnancy woman: woman who are submitted to elective Cesarean Section in spinal anesthesia
  Interventions: Diagnostic Test: B-Type natriuretic peptide (BNP) serum values; Device: Pulmonary echography; Other: urine collection

INTERVENTIONS:
Diagnostic Test: B-Type natriuretic peptide (BNP) serum values — evaluation BNP serum values:
  * pre- Cesarean Section (30 minutes before surgery)
  * post- Cesarean Section (6 hour and 24 hour after surgery)
Device: Pulmonary echography — Pulmonary echography:
  * pre- Cesarean Section (30 minutes before surgery)
  * post- Cesarean Section (6 hour and 24 hour after surgery)
Other: urine collection — 6 hour and 24 hour urine collection after Cesarean Section

SUMMARY:
Pregnancy is characterized by many biohumoral changes: circulation, respiratory mechanics, oncotic pressure, vascular permeability and many other systems are affected.

Vascular permeability is controlled by endothelial glycocalyx. Several factors such as sepsis, ischemia / reperfusion, inflammatory mediators, trauma, surgery including the Cesarean Section and fluid overload can increase vascular permeability due to a glycocalyx damage.

During Cesarean Section under subarachnoid anesthesia, hypotension may occur. It is a common side effect caused by reduced preload due to aortocaval compression by the uterus. Furthermore, subarachnoid anesthesia causes block of the sympathetic preganglionic fibers which is associated with vasodilation. These changes often require the use of vasopressors and fluids.

A fluid overload associated with the physiological and pathological factors discussed earlier might cause an increased risk of pulmonary edema and acute respiratory failure (IRA) in women undergoing cesarean section under arachnoid anesthesia.

IRA occurs in less than 0.2% of total pregnancies but it is one of the most common cause of admission to intensive care unit in pregnant women.

Among the causes that can lead to IRA in the last trimester of pregnancy we find pneumopathies such as asthma, pulmonary embolism due to amniotic fluid and pulmonary edema related to severe preeclampsia.

Diagnosis of pulmonary edema can be clinical or sub-clinical through laboratory tests such as BNP (b-type natriuretic peptide). It might also be necessary to execute instrumental examinations such as chest radiography (contraindicated in pregnancy) or trans-thoracic ultrasound.

Hypothesis: correlation between subarachnoid anesthesia, fluidic therapy and BNP values and ultrasound pattern

ELIGIBILITY:
Inclusion Criteria:

woman submit elective Cesarean Section:

* age > 18 years
* American Society of Anesthesiologists (ASA) physical status classification system > 2
* > 37 gestational age
* arterial pressure >/ = 140/90 mmHg and proteinuria < 300 mmHg during anesthesia pre-examination
* no known cardiovascular/respiratory disease
* pre-partum pulmonary echography

Exclusion Criteria:

* age < 18 years
* pulmonary echographic windows not satisfying
* blood loss during Cesarean Section more than 1000 mL and/or necessity to administer colloid
* postpartum hemorrhage within the first 24 hours following childbirth
* pre-eclamptic sign/symptoms within the first 5 days following childbirth
* twin pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients' anthropometric data were collected, data related to the anesthetic technique, pharmacological and intraoperative fluid therapy, sensory level reached after subarachnoid anesthesia, sensory level and motor blockade at discharge from the operating room. We also collected BNP serum values and pulmonary ultrasound images at 6 and 24 h after the intervention. Diuresis collection at 6 and 24 h after the intervention was registered as well as water balance.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-12-17 (Actual); Primary Completion 2018-08-08 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Ultrasound pulmonary variations | pulmonary echography is made 30 minutes before Cesarean Section, 6 and 24 hours after surgery
  The main goal of our study is to evaluate, preoperatively, the incidence of ultrasound pulmonary variations in pregnant women attending elective Cesarean Section

SECONDARY OUTCOMES:
subclinical pulmonary echography variation | pulmonary echography is made 30 minutes before Cesarean Section, 6 and 24 hours after surgery
  Evaluating the incidence of subclinical variations in ecographic lung characteristics at 6 and 24 hours after Cesarean Section
B-type natriuretic peptide serum value variation | B-type natriuretic peptide serum level is sampled 30 minutes before Cesarean Section, 6 and 24 hours after surgery 30 minutes before Cesarean Section, 6 and 24 hours after surgery
  Finding if there is any correlation between preoperative b-type natriuretic peptide and ecographic lung characteristics in pregnants, before and 24 hours after Cesarean Section
fluid administration and pulmonary echography variation | pulmonary echography is made 30 minutes before Cesarean Section, 6 and 24 hours after surgery
  Finding if there is any correlation between intraoperative fluids administered and ecographic lung characteristics

REFERENCES:
- [Background] Bamfo JE, Kametas NA, Nicolaides KH, Chambers JB. Maternal left ventricular diastolic and systolic long-axis function during normal pregnancy. Eur J Echocardiogr. 2007 Oct;8(5):360-8. doi: 10.1016/j.euje.2006.12.004. Epub 2007 Feb 23. PMID 17321800
- [Background] Campos O, Andrade JL, Bocanegra J, Ambrose JA, Carvalho AC, Harada K, Martinez EE. Physiologic multivalvular regurgitation during pregnancy: a longitudinal Doppler echocardiographic study. Int J Cardiol. 1993 Jul 15;40(3):265-72. doi: 10.1016/0167-5273(93)90010-e. PMID 8225661
- [Background] Lapinsky SE. Acute respiratory failure in pregnancy. Obstet Med. 2015 Sep;8(3):126-32. doi: 10.1177/1753495X15589223. Epub 2015 Jun 10. PMID 27512467
- [Background] Pereira A, Krieger BP. Pulmonary complications of pregnancy. Clin Chest Med. 2004 Jun;25(2):299-310. doi: 10.1016/j.ccm.2004.01.010. PMID 15099890
- [Background] Chappell D, Jacob M, Hofmann-Kiefer K, Conzen P, Rehm M. A rational approach to perioperative fluid management. Anesthesiology. 2008 Oct;109(4):723-40. doi: 10.1097/ALN.0b013e3181863117. PMID 18813052
- [Background] Resnik JL, Hong C, Resnik R, Kazanegra R, Beede J, Bhalla V, Maisel A. Evaluation of B-type natriuretic peptide (BNP) levels in normal and preeclamptic women. Am J Obstet Gynecol. 2005 Aug;193(2):450-4. doi: 10.1016/j.ajog.2004.12.006. PMID 16098869